CLINICAL TRIAL: NCT00395798
Title: Effect of Conservative Treatment With Cervical Collar in Patients With Cervical Radiculopathy and Radicular Pain. A Randomized Controlled Study
Brief Title: Effect of Cervical Collar in Cervical Radicular Pain.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Collaborators: Norwegian Fund for Postgraduate Training in Physiotherapy (Other)
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EVisi
Record Dates: First submitted 2006-11-02; First posted 2006-11-03 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2006-05

CONDITIONS: Cervical Radicular Pain
Keywords: cervical intervertebral disc displacement; cervical spondylosis; radiculopathy; neck collar; brace; physiotherapy; treatment; rehabilitation
MeSH Terms: conditions — Spondylosis; Radiculopathy

INTERVENTIONS:
Device: Soft or stiff cervical collar(device), neck school(behavior)

SUMMARY:
Objectives:The purpose of this study is to determine if use of nech collar (stiff or soft)will improve the possibility to obtain painrelief in patients with cervical radicular pain. We will compare short term (six weeks and three months) and long term ( one year) effect of six weeks use of neck collar (stiff or soft)together with "neck school information" with "neck school information" alone.

ELIGIBILITY:
Inclusion Criteria:

* cervical radicular pain caused by herniated disc og spondolytic spurs
* written consent from patient

Exclusion Criteria:

* previous necksurgery
* whiplash or other necktrauma
* serious diseases somatic or psychiatric
* patients not able to speak and read Norwegian well
* insufficient correlation between clinical and radiological findings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2004-01; Study Completion 2007-08

PRIMARY OUTCOMES:
painscore on visual analog scale 0-100mm after 6weeks treatment

SECONDARY OUTCOMES:
painscore visual analog scale 0-100mm after 3weeks,3months,1year
Functional status on Neck pain and disability index after 3weeks,6weeks,3months,1 year
Quality of life score, Cantrils Ladder Scale 3 weeks,6weeks,3 months,1 year

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Graver, PhD, Study Director — Ullevaal University Hospital
Locations (1):
- Ullevaal University Hospital, Oslo, Norway